CLINICAL TRIAL: NCT06631807
Title: The Impact of the Years of Blindness on Sleep and Dreaming Processes and Possible Relationships With Spatial Abilities
Brief Title: The Impact of the Years of Blindness on Sleep and Dreaming Processes and the Relationships With Spatial Abilities
Status: Enrolling by invitation | Type: Observational
Sponsor: Istituto Italiano di Tecnologia (Other)
Responsible Party: Sponsor
Other Study IDs: IIT_UVIP_BLINDREAM_2022
Record Dates: First submitted 2024-08-31; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Blindness; Visual Impairment
Keywords: Blindness; sleep; PSG; circadian; dream; spatial abilities
MeSH Terms: conditions — Blindness; Vision Disorders; Spatial Navigation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Salivary sample for melatonin analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Blind and severely visually impaired (BSI): This group is composed of adults participants (ages of ≥ 18 and ≤ 85 years) with an impairment of the peripheral visual system (i.e., involving pre-chiasmatic structures, such as the retina and optic nerve). The visual deficit can be congenital (from birth) or have a late onset. Participants with visual impairment, classified according to the current diagnostic criteria, must have residual vision lower than 1.0 LogMAR. Participant of any gender and ethnicity are considered, provided they have a good knowledge of the Italian language.
- Control: Control group is composed of adult participants (without visual deficits) age and gender matched with the BSI group.

SUMMARY:
This study aims to assess the impact of blindness on sleep and dreaming processes and the relationship with spatial perceptual performance, examining the link with clinical and psychological indices, neurobiological features, and electrophysiological measures.

DETAILED DESCRIPTION:
BLINDREAM is an observational neuropsychology study purely for scientific purposes, with no diagnostic or therapeutic aims. This study aims to assess the impact of blindness on sleep and dream processes and their relationship with perceptual and spatial memory performance, examining the connection with clinical, psychological/behavioral indices, neurobiological characteristics, and electrophysiological measures. Specifically, the study seeks to test the following hypotheses:

* Circadian Rhythm Desynchronization: To determine if visual deprivation leads to circadian rhythm desynchronization in both congenitally blind individuals and those with late-onset blindness after many years of visual deprivation. Specifically, whether greater circadian desynchronization is associated with poorer performance in perceptual and spatial memory tasks in blind subjects.
* Sleep Structure: To investigate if circadian desynchronization affects sleep structure in blind individuals and if it is the sole factor influencing sleep structure. We hypothesize that even blind subjects with a normally modulated circadian rhythm due to the light-dark cycle show significant differences from sighted controls, particularly in terms of sleep microstructure (figures) and macrostructure (stages) involved in sensorimotor processing and spatial information consolidation.
* Dream Recall and Spatial Abilities: To examine if there is a significant difference in dream recall frequency and specific spatial tasks between the two groups. Specifically, whether a higher presence of visual content in dreams predicts better spatial skills, and whether increased eye movement in dreams correlates with better spatial abilities in blind subjects.

These findings will enable initial assessments that may lead to the development of new tools and rehabilitation protocols for blind individuals.

The study will be conducted in three experimental phases over a total of one week per participant:

* Phase 1: Sleep and Dream Assessment: This includes two measures-1A. Questionnaires and 1B. Polysomnography.
* Phase 2: Circadian Assessment: This includes three measures-2A. Actigraphy (worn for one week), 2B. Salivary melatonin analysis, and 2C. Dream diary.
* Phase 3: Neuropsychological Assessment: This involves evaluating several conditions with two specific configurations-3A. Assessment of spatial perceptual functions and 3B. Assessment of spatial memory.

Each phase involves different sessions: the circadian assessment requires wearing an actigraphic bracelet for a week, during which salivary melatonin will also be measured; the sleep and dream assessment involves wearing a home polysomnograph for one night and completing a verbal dream diary for one week; and the neuropsychological assessment will be conducted in a single session lasting between approximately 30 minutes and 2 hours.

The study will include adult individuals both with and without visual impairments. The visual impairment may be congenital or acquired later in life. Control group participants will be selected to match the experimental group (those with visual impairments) in terms of age and gender. Due to the proof-of-concept nature of the study and the lack of prior estimates of effect sizes, power calculations are not currently possible. The sample size is therefore based on a provisional and conservative estimate of recruitment capacity, informed by previous literature. However, efforts will be made to conduct interim analyses to estimate effect sizes based on the primary outcome and adjust assumptions accordingly. The study currently aims to recruit 20 blind participants and 20 healthy controls.

Therefore, the preliminary data will utilize the Power Analysis method to calculate the minimum sample size required to achieve a correct effect size for a given dimension. The data will be analyzed using both parametric and non-parametric tests, and differences between groups will be assessed with t-tests, ANOVA, TANCOVA, and linear mixed models where appropriate. An appropriate post-hoc test will be conducted if significance is found. The significance level will be considered at p<0.05. Where necessary, parametric techniques will be replaced by non-parametric equivalents. The standard software used will include: Matlab, R, Origin, Statistica, and SPSS, recognized in the research field. For the analysis of electroencephalographic data, EEGlab and/or Fieldtrip toolboxes will be utilized.

ELIGIBILITY:
Inclusion Criteria:

* Signature of the informed consent;
* The participating subjects may have typical or atypical development (i.e., group with visual disability). In the case of visual impairment, the disability should be congenital (from birth) or late onset. Furthermore, the following requirements must be met: subjects with visual disabilities must be classified according to current diagnostic rules, with visual problems present from birth or occurring later, with residual vision lower than 1.3 LogMAR;
* Age range required is ≥ 18 years old and ≤ 85 years old;
* Any Gender;
* Any ethnicity, as long as a good knowledge of the Italian language.

Exclusion Criteria:

* Participant with a disability/condition/comorbidity that prevents participation and/or does not guarantee the safety of the patient during the execution of the tests and/or does not guarantee the quality/reliability of the data:

  * Tactile and/or acoustic hypersensitivity (specifically, the tolerance of the equipment will be assessed);
  * Deafness;
  * Taking drugs and neuroactive substances and having taken them in the last six months;
  * Comorbidity with another clinically significant and uncontrolled pathology;
  * Being affected, to the best of their knowledge, by pathologies of the central nervous system, and having suffered from epileptic episodes, even minor ones, and convulsive crises in general;
  * Being affected, to the best of their knowledge, by cardio-respiratory pathologies that can influence the macro and microstructure of sleep.
* Lack of signature of consent or incomplete consent to acknowledge the incompatibilities for participation in the study;
* To the best of their knowledge, IQ values lower than the threshold limit of normality according to one of the recognized international scales.
* Pregnant women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include adult individuals both with and without visual impairments. The visual impairment may be congenital or acquired later in life. Control group participants will be selected to match the experimental group (those with visual impairments) in terms of age and gender. Due to the proof-of-concept nature of the study and the lack of prior estimates of effect sizes, power calculations are not currently possible. The sample size is therefore based on a provisional and conservative estimate of recruitment capacity, informed by previous literature. However, efforts will be made to conduct interim analyses to estimate effect sizes based on the primary outcome and adjust assumptions accordingly. The study currently aims to recruit 20 blind participants and 20 healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-10-04 (Estimated); Study Completion 2025-10-04 (Estimated)

PRIMARY OUTCOMES:
Sleep macrostructure | Through study completion, an average of 18 months
  Percentage of sleep stages and spectrogram
Sleep microstructure | Through study completion, an average of 18 months
  Analysis of sleep spindles
Sleep microstructure | Through study completion, an average of 18 months
  Analysis of slow waves
Sleep quality - PSQI | Through study completion, an average of 12 months
  Pittsburgh Sleep Quality Index. The seven component scores are then summed to yield a global PSQI score, which has a range of 0-21; higher scores indicate worse sleep quality.
Sleep Quality - questionnaire to predict N24HSWD | Through study completion, an average of 12 months
  Pre-Screening questionnaire to predict Non-24-hours sleep-wake disorders. The questionnaire assesses sleep-wake patterns, focusing on irregularities such as difficulty maintaining a regular sleep schedule and daytime dysfunction. It includes a set of eight key questions.
  The scoring system can yield final values greater than or less than zero:
  1. Values greater than zero suggest that the patient should be evaluated for N24HSWD.
  2. Values less than zero indicate the need for assessment for other sleep disorders.
  This tool serves as an initial filter, guiding whether further diagnostic measures, like actigraphy or melatonin rhythm analysis, are necessary
Sleep quality - MEQ | Through study completion, an average of 12 months
  Morningness -Eveningness Questionnaire. It is a Self-reported assessment of morningness and eveningness preferences with a 19 multiple choice items (4-5 point numerical scale). The sum gives a score ranging from 16 to 86; scores of 41 and below indicate "evening types", scores of 59 and above indicate "morning types", scores between 42-58 indicate "intermediate types".
Circadian shift | Through study completion, an average of 18 months
  Melatonin sample ELISA protocol
Circadian shift | Through study completion, an average of 18 months
  Actigraphy measures
Spatial perception ability | Through study completion, an average of 12 months
  Spatial and temporal bisection
Spatial memory ability | Through study completion, an average of 12 months
  Audiocorsi
Dream content evaluation - DRFS | Through study completion, an average of 12 months
  The Dream Recall Frequency Scale (DRFS) is a useful tool for assessing how often individuals remember their dreams. This scale can help distinguish between high dreamers (those who frequently recall dreams) and low dreamers (those who rarely remember dreams). The scale typically ranges from 0 to 5, where a higher value indicates more frequent recall of dreams.
Dream content evaluation - VDAS | Through study completion, an average of 12 months
  The Van Dream Anxiety Scale (VDAS) is a tool used to assess the severity of nightmares and dream anxiety. The VDAS consists of a set of items that measure the frequency, intensity, and emotional impact of nightmares, as well as their interference with daily functioning. The scale typically provides a range of scores from 0 to 68, where. Higher scores indicate greater severity of nightmares and dream-related anxiety.
Dream content evaluation | Through study completion, an average of 18 months
  Dream Diary

CONTACTS AND LOCATIONS:
Locations (1):
- U.O. Clinica Neurologica Ambul. disturbi del sonno ed epilessia; IRCCS Ospedale Policlinico San Martino, Genova, Italy

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication

REFERENCES:
- [Result] Hartley S, Dauvilliers Y, Quera-Salva MA. Circadian Rhythm Disturbances in the Blind. Curr Neurol Neurosci Rep. 2018 Aug 6;18(10):65. doi: 10.1007/s11910-018-0876-9. PMID 30083814
- [Result] Lockley SW, Skene DJ, Butler LJ, Arendt J. Sleep and activity rhythms are related to circadian phase in the blind. Sleep. 1999 Aug 1;22(5):616-23. doi: 10.1093/sleep/22.5.616. PMID 10450596
- [Result] Depner CM, Stothard ER, Wright KP Jr. Metabolic consequences of sleep and circadian disorders. Curr Diab Rep. 2014 Jul;14(7):507. doi: 10.1007/s11892-014-0507-z. PMID 24816752
- [Result] Lockley SW, Dijk DJ, Kosti O, Skene DJ, Arendt J. Alertness, mood and performance rhythm disturbances associated with circadian sleep disorders in the blind. J Sleep Res. 2008 Jun;17(2):207-16. doi: 10.1111/j.1365-2869.2008.00656.x. PMID 18482109
- [Result] Aubin S, Christensen JAE, Jennum P, Nielsen T, Kupers R, Ptito M. Preserved sleep microstructure in blind individuals. Sleep Med. 2018 Feb;42:21-30. doi: 10.1016/j.sleep.2017.11.1135. Epub 2017 Dec 7. PMID 29458742
- [Result] Christensen JAE, Aubin S, Nielsen T, Ptito M, Kupers R, Jennum P. Rapid eye movements are reduced in blind individuals. J Sleep Res. 2019 Dec;28(6):e12866. doi: 10.1111/jsr.12866. Epub 2019 Apr 26. PMID 31025801
- [Result] Meaidi A, Jennum P, Ptito M, Kupers R. The sensory construction of dreams and nightmare frequency in congenitally blind and late blind individuals. Sleep Med. 2014 May;15(5):586-95. doi: 10.1016/j.sleep.2013.12.008. Epub 2014 Feb 18. PMID 24709309
- [Result] Chellappa SL, Cajochen C. Ultradian and circadian modulation of dream recall: EEG correlates and age effects. Int J Psychophysiol. 2013 Aug;89(2):165-70. doi: 10.1016/j.ijpsycho.2013.03.006. Epub 2013 Mar 20. PMID 23524011
- [Result] Wamsley EJ, Tucker M, Payne JD, Benavides JA, Stickgold R. Dreaming of a learning task is associated with enhanced sleep-dependent memory consolidation. Curr Biol. 2010 May 11;20(9):850-5. doi: 10.1016/j.cub.2010.03.027. Epub 2010 Apr 22. PMID 20417102
- [Result] Picard-Deland C, Aumont T, Samson-Richer A, Paquette T, Nielsen T. Whole-body procedural learning benefits from targeted memory reactivation in REM sleep and task-related dreaming. Neurobiol Learn Mem. 2021 Sep;183:107460. doi: 10.1016/j.nlm.2021.107460. Epub 2021 May 18. PMID 34015442
- [Result] Eichenlaub JB, Bertrand O, Morlet D, Ruby P. Brain reactivity differentiates subjects with high and low dream recall frequencies during both sleep and wakefulness. Cereb Cortex. 2014 May;24(5):1206-15. doi: 10.1093/cercor/bhs388. Epub 2013 Jan 2. PMID 23283685
- [Result] Borbely AA, Daan S, Wirz-Justice A, Deboer T. The two-process model of sleep regulation: a reappraisal. J Sleep Res. 2016 Apr;25(2):131-43. doi: 10.1111/jsr.12371. Epub 2016 Jan 14. PMID 26762182
- [Result] Dirks C, Grunewald D, Young P, Heidbreder A. [Pilot study to investigate sleep disorders in the blind and persons with relevant visual impairment]. Ophthalmologe. 2019 May;116(5):435-440. doi: 10.1007/s00347-018-0723-z. German. PMID 29789897
- [Result] Lewy AJ, Newsome DA. Different types of melatonin circadian secretory rhythms in some blind subjects. J Clin Endocrinol Metab. 1983 Jun;56(6):1103-7. doi: 10.1210/jcem-56-6-1103. PMID 6841552
- [Result] De Volder AG, Toyama H, Kimura Y, Kiyosawa M, Nakano H, Vanlierde A, Wanet-Defalque MC, Mishina M, Oda K, Ishiwata K, Senda M. Auditory triggered mental imagery of shape involves visual association areas in early blind humans. Neuroimage. 2001 Jul;14(1 Pt 1):129-39. doi: 10.1006/nimg.2001.0782. PMID 11525322
- [Result] Richardson C, Micic G, Cain N, Bartel K, Maddock B, Gradisar M. Cognitive performance in adolescents with Delayed Sleep-Wake Phase Disorder: Treatment effects and a comparison with good sleepers. J Adolesc. 2018 Jun;65:72-84. doi: 10.1016/j.adolescence.2018.03.002. Epub 2018 Mar 16. PMID 29555485
- [Result] Chellappa SL, Morris CJ, Scheer FAJL. Circadian misalignment increases mood vulnerability in simulated shift work. Sci Rep. 2020 Oct 29;10(1):18614. doi: 10.1038/s41598-020-75245-9. PMID 33122670
- [Result] Le Bon O. Relationships between REM and NREM in the NREM-REM sleep cycle: a review on competing concepts. Sleep Med. 2020 Jun;70:6-16. doi: 10.1016/j.sleep.2020.02.004. Epub 2020 Feb 15. PMID 32179430
- [Result] Aubin S, Jennum P, Nielsen T, Kupers R, Ptito M. Sleep structure in blindness is influenced by circadian desynchrony. J Sleep Res. 2018 Feb;27(1):120-128. doi: 10.1111/jsr.12548. Epub 2017 Jun 16. PMID 28621018
- [Result] Leger D, Guilleminault C, Santos C, Paillard M. Sleep/wake cycles in the dark: sleep recorded by polysomnography in 26 totally blind subjects compared to controls. Clin Neurophysiol. 2002 Oct;113(10):1607-14. doi: 10.1016/s1388-2457(02)00221-3. PMID 12350437
- [Result] Hono T, Hiroshige Y, Miyata Y. A case report on EEG nocturnal sleep in visually impaired persons aged in their 30s and 50s. Psychiatry Clin Neurosci. 1999 Apr;53(2):145-7. doi: 10.1046/j.1440-1819.1999.00501.x. PMID 10459673
- [Result] Scrofani A, Cioni M, Filetti S, Lanaia F, Pennisi G, Bella R, Grasso A. Changes in sleep spindle activity of subject with chronic somatosensitive and sensorial deficits. Preliminary results. Ital J Neurol Sci. 1996 Dec;17(6):423-8. doi: 10.1007/BF01997717. PMID 8978449
- [Result] Kerr NH, Foulkes D, Schmidt M. The structure of laboratory dream reports in blind and sighted subjects. J Nerv Ment Dis. 1982 May;170(5):286-94. doi: 10.1097/00005053-198205000-00006. No abstract available. PMID 7069416
- [Result] Bertolo H, Paiva T, Pessoa L, Mestre T, Marques R, Santos R. Visual dream content, graphical representation and EEG alpha activity in congenitally blind subjects. Brain Res Cogn Brain Res. 2003 Feb;15(3):277-84. doi: 10.1016/s0926-6410(02)00199-4. PMID 12527101
- [Result] Sabo KT, Kirtley DD. Emotions in the dreams of the blind. Int J Rehabil Res. 1980;3(3):382-5. doi: 10.1097/00004356-198009000-00013. No abstract available. PMID 7450997
- [Result] Gori M. Multisensory Integration and Calibration in Children and Adults with and without Sensory and Motor Disabilities. Multisens Res. 2015;28(1-2):71-99. doi: 10.1163/22134808-00002478. PMID 26152053
- [Result] Gori M, Sandini G, Burr D. Development of visuo-auditory integration in space and time. Front Integr Neurosci. 2012 Sep 17;6:77. doi: 10.3389/fnint.2012.00077. eCollection 2012. PMID 23060759
- [Result] Gori M, Del Viva M, Sandini G, Burr DC. Young children do not integrate visual and haptic form information. Curr Biol. 2008 May 6;18(9):694-8. doi: 10.1016/j.cub.2008.04.036. PMID 18450446
- [Result] Gori M, Sandini G, Martinoli C, Burr D. Poor haptic orientation discrimination in nonsighted children may reflect disruption of cross-sensory calibration. Curr Biol. 2010 Feb 9;20(3):223-5. doi: 10.1016/j.cub.2009.11.069. Epub 2010 Jan 28. PMID 20116249
- [Result] Roder B, Rosler F, Spence C. Early vision impairs tactile perception in the blind. Curr Biol. 2004 Jan 20;14(2):121-4. PMID 14738733
- [Result] Zwiers MP, Van Opstal AJ, Cruysberg JR. A spatial hearing deficit in early-blind humans. J Neurosci. 2001 May 1;21(9):RC142: 1-5. doi: 10.1523/JNEUROSCI.21-09-j0002.2001. PMID 11312316
- [Result] Cappagli G, Cocchi E, Gori M. Auditory and proprioceptive spatial impairments in blind children and adults. Dev Sci. 2017 May;20(3). doi: 10.1111/desc.12374. Epub 2015 Nov 27. PMID 26613827
- [Result] Gori M, Sandini G, Martinoli C, Burr DC. Impairment of auditory spatial localization in congenitally blind human subjects. Brain. 2014 Jan;137(Pt 1):288-93. doi: 10.1093/brain/awt311. Epub 2013 Nov 21. PMID 24271326
- [Result] Gori M, Amadeo MB, Campus C. Temporal cues trick the visual and auditory cortices mimicking spatial cues in blind individuals. Hum Brain Mapp. 2020 Jun 1;41(8):2077-2091. doi: 10.1002/hbm.24931. Epub 2020 Feb 12. PMID 32048380
- [Result] Amadeo MB, Campus C, Gori M. Years of Blindness Lead to "Visualize" Space Through Time. Front Neurosci. 2020 Aug 4;14:812. doi: 10.3389/fnins.2020.00812. eCollection 2020. PMID 32848573
- [Result] Gori M, Amadeo MB, Campus C. Temporal Cues Influence Space Estimations in Visually Impaired Individuals. iScience. 2018 Aug 31;6:319-326. doi: 10.1016/j.isci.2018.07.003. Epub 2018 Aug 1. PMID 30240622
- [Result] Setti W, Cuturi LF, Engel I, Picinali L, Gori M. The influence of early visual deprivation on audio-spatial working memory. Neuropsychology. 2022 Jan;36(1):55-63. doi: 10.1037/neu0000776. Epub 2021 Oct 14. PMID 34647755
- [Result] Setti W, Cuturi LF, Cocchi E, Gori M. A novel paradigm to study spatial memory skills in blind individuals through the auditory modality. Sci Rep. 2018 Sep 6;8(1):13393. doi: 10.1038/s41598-018-31588-y. PMID 30190584
- [Result] Ruggiero G, Iachini T. The role of vision in the Corsi block-tapping task: evidence from blind and sighted people. Neuropsychology. 2010 Sep;24(5):674-9. doi: 10.1037/a0019594. PMID 20804256
- [Result] Vecchi T, Tinti C, Cornoldi C. Spatial memory and integration processes in congenital blindness. Neuroreport. 2004 Dec 22;15(18):2787-90. PMID 15597055
- [Result] Aubin S, Gacon C, Jennum P, Ptito M, Kupers R. Altered sleep-wake patterns in blindness: a combined actigraphy and psychometric study. Sleep Med. 2016 Aug;24:100-108. doi: 10.1016/j.sleep.2016.07.021. Epub 2016 Aug 31. PMID 27810175
- [Result] Flynn-Evans EE, Lockley SW. A Pre-Screening Questionnaire to Predict Non-24-Hour Sleep-Wake Rhythm Disorder (N24HSWD) among the Blind. J Clin Sleep Med. 2016 May 15;12(5):703-10. doi: 10.5664/jcsm.5800. PMID 26951421
- [Result] Schredl M. Reliability and stability of a dream recall frequency scale. Percept Mot Skills. 2004 Jun;98(3 Pt 2):1422-6. doi: 10.2466/pms.98.3c.1422-1426. PMID 15291233